CLINICAL TRIAL: NCT04869410
Title: Accuracy of Broselow Tape and Cole Formulation in Predicting Uncuffed Endotracheal Tube Size in Pediatric Patients
Brief Title: Comparison of Modified Broselow Tape and Cole Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IndonesiaUAnes103
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Predicting Uncuffed Endotracheal Tube Size in Pediatric Anesthesia
Keywords: Uncuffed endotracheal tube; Pediatric; Cole Formula; Broselow Tape

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broselow Tape (Active Comparator): Patient will given an intubation using uncuffed endotracheal tube size based on Modified Broselow Tape
  Interventions: Procedure: Modification Broselow Tape; Procedure: Cole Formula
- Cole Formula (Active Comparator): Patient will given an intubation using uncuffed endotracheal tube size based on Cole Formula
  Interventions: Procedure: Modification Broselow Tape; Procedure: Cole Formula

INTERVENTIONS:
Procedure: Modification Broselow Tape — Intubation using modified Broselow Tape prediction for predicting ETT size
Procedure: Cole Formula — Intubation using Cole Formula prediction for predicting ETT size

SUMMARY:
This study aimed to determine the accuracy of modified Broselow tape measurements compared to Cole formula in predicting the size of uncuffed endotracheal tubes in Indonesian pediatrics

DETAILED DESCRIPTION:
110 subjects were given informed consent before enrolling the study and randomized into two groups, modified Broselow Tape and Cole formula. Preoperatively, prediction of suitable ETT size was performed based on Cole formula and Modified Broselow Tape. In the operating theatre, general anesthesia induction was performed with sevoflurane 4-8 vol%, fentanyl 2 μcg/kg BW, and atracurium 0.5 mg/kg BW. Laryngoscopy was performed, and an uncuffed polyvinyl chloride endotracheal tubes, whose size was based on the Cole formula, was inserted. An appropriate size of the endotracheal tube was confirmed if the endotracheal tube could go through the cricoid ring smoothly, and no air leakage found when ventilating with an inspiratory pressure of 15-20 cmH2O. The surgery and anesthesia would proceed if the correct size of the endotracheal tube were successfully inserted. If the tube couldn't pass the cricoid smoothly or air leakage was found when ventilated with an inspiratory pressure of 15-20 cmH2O, the endotracheal tube should be replaced with a bigger or smaller size.

ELIGIBILITY:
Inclusion Criteria:

* pediatrics aged 1 - 6 y o
* ASA I-II
* patients went through elective surgery with Genaral anesthesia
* Need to intubated with uncuffed ETT

Exclusion Criteria:

* patients with growth and development disorders
* patients whom height that was out of range in modified Broselow tape
* patients with possible airway difficulty or obstruction
* patients with respiratory diseases, underweight and obese

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Appropriate size of uncuffed endotracheal tube | before procedure
  endotracheal tube could go through the cricoid ring smoothly, and no air leakage found when ventilating with an inspiratory pressure of 15-20 cmH2O

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospotal, Jakarta Pusat, DKI Jaka, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hofer CK, Ganter M, Tucci M, Klaghofer R, Zollinger A. How reliable is length-based determination of body weight and tracheal tube size in the paediatric age group? The Broselow tape reconsidered. Br J Anaesth. 2002 Feb;88(2):283-5. doi: 10.1093/bja/88.2.283. PMID 11878662
- [Background] Park HP. Appropriate tube size selection based on radiological images. Korean J Anesthesiol. 2014 Mar;66(3):181-2. doi: 10.4097/kjae.2014.66.3.181. No abstract available. PMID 24729837
- [Background] Schramm C, Knop J, Jensen K, Plaschke K. Role of ultrasound compared to age-related formulas for uncuffed endotracheal intubation in a pediatric population. Paediatr Anaesth. 2012 Aug;22(8):781-6. doi: 10.1111/j.1460-9592.2012.03889.x. Epub 2012 May 21. PMID 22612446
- [Background] Jang HY, Shin SD, Kwak YH. Can the Broselow tape be used to estimate weight and endotracheal tube size in Korean children? Acad Emerg Med. 2007 May;14(5):489-91. doi: 10.1197/j.aem.2006.12.014. Epub 2007 Mar 23. PMID 17384410
- [Result] Shih MH, Chung CY, Su BC, Hung CT, Wong SY, Wong TK. Accuracy of a new body length-based formula for predicting tracheal tube size in Chinese children. Chang Gung Med J. 2008 May-Jun;31(3):276-80. PMID 18782950